CLINICAL TRIAL: NCT01452152
Title: Pharmacogenomics of Anti-platelet Intervention-2 (PAPI-2) Study: A Prospective, Multicenter, Randomized Trial of Genotype-directed (G-D)Versus Standard of Care (SOC)Anti-platelet Therapy
Brief Title: Pharmacogenomics of Anti-platelet Intervention-2 (PAPI-2) Study
Acronym: PAPI-2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated by study sponsor.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alan Shuldiner, Professor, School of Medicine; Head, Division of Endocrinology, Diabetes and Nutrition, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00047385; 9U01HL105198-06 (NIH)
Record Dates: First submitted 2011-10-10; First posted 2011-10-14 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Diseases; Acute Coronary Syndrome
Keywords: Pharmacogenomics; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome | interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Genotype-directed, clopidogrel (Experimental): Participants randomized to the G-D group will have CYP2C19 genotype analysis performed. CYP2C19 extensive and ultrarapid metabolizers will receive clopidogrel.
  Interventions: Drug: clopidogrel
- Genotype-directed, prasugrel (Experimental): Participants randomized to the G-D group will have CYP2C19 genotype analysis performed. CYP2C19 intermediate and poor metabolizers will receive prasugrel.
  Interventions: Drug: prasugrel
- Standard of Care (No Intervention): Participants randomized to the SOC group will not have CYP2C19 genotype analysis performed. They will receive dual anti-platelet therapy guided by the judgment of their treating physician according to standard medical practice irrespective of genotype.

INTERVENTIONS:
Drug: clopidogrel — clopidogrel 75 mg/day plus aspirin 81-162 mg/day for one year
  Other Names: Plavix
  Arms: Genotype-directed, clopidogrel
Drug: prasugrel — Prasugrel 5-10 mg/day plus aspirin 81-162 mg/day for one year
  Other Names: Effient
  Arms: Genotype-directed, prasugrel

SUMMARY:
It is standard treatment to take anti-platelet medication after cardiac catheterization and stent placement to help prevent the formation of blood clots that may cause heart attack or stroke. The most commonly used anti-platelet medicine is clopidogrel (Plavix®). However, researchers have found that people vary in their response to clopidogrel, in part because of differences in their genes. Prasugrel (Effient®)is another anti-platelet medication used to prevent clots. The genetic differences that affect clopidogrel response do not affect prasugrel response. Recently, the FDA added a warning to the label of clopidogrel to notify doctors and patients with certain genetic differences may not get the full benefit from clopidogrel. Despite this, genetic testing for these variations is not usually done in standard medical practice. The purpose of this study is to see if patients with certain gene differences have fewer major cardiac events after stent placement if they are given anti-platelet therapy guided by their individual genetic type compared to standard anti-platelet therapy.

DETAILED DESCRIPTION:
Over a three-year period, a total of 7,200 patients undergoing percutaneous coronary intervention (PCI) in whom dual anti-platelet therapy is indicated for at least one year and meet the eligibility criteria, will be recruited from five or more clinical sites. Patients presenting to the cardiac clinics, emergency departments, catheterization laboratories, and other acute care units (e.g. CCU) who will have coronary angiography or have had angiography and PCI will be offered participation. Following informed consent, patients will have baseline data and specimens collected, and eligibility confirmed. Patients will be randomized in equal numbers to the G-D arm or SOC arm. Immediately following randomization, a blood sample from patients assigned to the G-D arm will be sent for CYP2C19 genotype analysis. Upon receipt of CYP2C19 genotype results, patients randomized to the G-D arm with the CYP2C19 *1/*1 genotype (extensive metabolizers) and *1/*17, and *17/*17 genotypes (ultrarapid metabolizers) will receive clopidogrel 75 mg/day plus aspirin 81-162 mg/day (group a). Those with *1/*2, *1/*3, *2/*17, and *3/*17 genotypes (intermediate metabolizers) and those with *2/*2, *2/*3, and *3/*3 genotypes (poor metabolizers) will receive prasugrel 5-10 mg/day plus aspirin 81-162 mg/day (group b). Patients randomized to the SOC arm will not be genotyped prospectively. They will receive dual anti-platelet therapy guided by the judgment of their treating physician according to standard medical practice irrespective of genotype (group c). Optionally, a subgroup of patients will return at 10 days after the randomization visit for platelet aggregation studies.

If our hypothesis is correct, i.e., that in intermediate and poor metabolizers, G-D anti-platelet therapy results in fewer cardiovascular events and has less or equivalent bleeding complications compared to SOC therapy, and is cost effective, this prospective randomized clinical trial will provide the evidence base to implement genotype-directed anti-platelet treatment algorithms broadly into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females between the ages of 20 and 74 years, inclusive
* Not more than four days post-PCI (percutaneous coronary intervention) with placement of one or more drug eluting or bare metal stents
* One or more stent(s) delivered with final TIMI 3 flow (thrombolysis in myocardial infarction grade 3) in the stented vessel(s)
* Must have evidence of one of the following:

  1. Three vessel disease;
  2. Two vessel disease with one of the following: estimated creatinine clearance <60, prior myocardial infarction, diabetes mellitus on treatment, peripheral artery disease, cerebrovascular disease, bifurcation stent, overlapping stents, or total stent deployment length > 40 mm in length;
  3. Single vessel disease with two of the following: estimated creatinine clearance <60, prior myocardial infarction, diabetes mellitus on treatment, peripheral artery disease, cerebrovascular disease, bifurcating stenting, overlapping stents, or total stent deployment length > 40 mm in length.
* Patients with acute MI (myocardial infarction) preceding the PCI must have CK-MB (bound combination of creatine kinase M and creatine kinase B) value lower than the prior value, before randomization
* Patients with peri-procedural MI, defined by CK-MB three times greater than upper reference limit (URL), must have CK-MB value lower than the prior value, before randomization. Peri-procedural MI will be screened per clinical suspicion.
* Have an indication for one year of dual anti-platelet therapy with a P2Y12 inhibitor and aspirin
* Agreement of the treating physician to prescribe anti-platelet therapy according to randomization and study dosing algorithm
* Ability to understand and comply with planned study procedures
* Provide written informed consent prior to study entry
* Agrees to authorize the collection and release of his/her medical information for the duration of the trial or until the subject withdraws

Exclusion Criteria:

* History of a gastrointestinal bleed within three months or a major, life threatening bleeding event (e.g., sub-arachnoid or intracranial hemorrhage)
* Active pathological bleeding (e.g. GI bleeding)
* History of bleeding diathesis or coagulopathy
* History of stroke or transient ischemic attack (TIA)
* Non-cardiac surgery within the prior 3 months
* Planned cardiac or non-cardiac surgery within the next 12 months
* CYP2C19 genotype already known to subject or research team from prior genetic testing
* Post-PCI CABG (coronary artery bypass graft) before randomization
* Planned warfarin or dabigatran therapy any time during the study period
* Known allergy to aspirin, clopidogrel or prasugrel
* Platelet count <100,000/mm3
* Hematocrit < 25%
* Pregnancy
* Concurrent enrollment in another trial that involves an investigational stent, antithrombotic or anti-platelet agent
* Any condition that would, in the opinion of the site investigator, place them at an unacceptable risk or render them unable to meet the requirements of the protocol
* Any subject, in the opinion of the investigator, not expected to tolerate or be adherent with one year of dual antiplatelet therapy

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Shuldiner, M.D., Principal Investigator — University of Maryland
Locations (5):
- United States (5):
  - Christiana Care Health System, Newark, Delaware
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Sinai Center for Thrombosis Research, Baltimore, Maryland
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Geisinger Health System, Danville, Pennsylvania

REFERENCES:
- [Background] Shuldiner AR, O'Connell JR, Bliden KP, Gandhi A, Ryan K, Horenstein RB, Damcott CM, Pakyz R, Tantry US, Gibson Q, Pollin TI, Post W, Parsa A, Mitchell BD, Faraday N, Herzog W, Gurbel PA. Association of cytochrome P450 2C19 genotype with the antiplatelet effect and clinical efficacy of clopidogrel therapy. JAMA. 2009 Aug 26;302(8):849-57. doi: 10.1001/jama.2009.1232. PMID 19706858

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Genotype-directed, Clopidogrel | Genotype-directed, Prasugrel | Standard of Care
Started | 5 | 0 | 4
Completed | 0 | 0 | 0
Not Completed | 5 | 0 | 4
Not completed — Study termination by sponsor | 5 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genotype-directed, Clopidogrel | Genotype-directed, Prasugrel | Standard of Care | Total
Number analyzed (Participants) | 5 | 0 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 | 0
  Between 18 and 65 years | 3 |  | 3 | 6
  >=65 years | 2 |  | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 2 | 3
  Male | 4 |  | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 1 | 1
  Not Hispanic or Latino | 5 |  | 3 | 8
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 1 | 1
  White | 5 |  | 2 | 7
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Post-randomization Cardiovascular Events
Description: Cardiovascular events include non-fatal myocardial infarction, non-fatal stroke, definite or probable stent thrombosis (ARC definition) and death secondary to any cardiovascular cause.
Time Frame: One year
Population: Zero participants were assigned to genotype-directed, prasugrel group
Measure: Number; unit: participants
Arm/Group | Genotype-directed, Clopidogrel | Genotype-directed, Prasugrel | Standard of Care
Number analyzed (Participants) | 5 | 0 | 4
participants | 0 |  | 0

2. Secondary Outcome: Occurrence of Bleeding Events
Description: Bleeding events will classified by the Bleeding Academic Research Consortium definition. The number of bleeding events will be tabulated.
Time Frame: One year
Population: Zero participants were assigned to genotype-directed, prasugrel group
Measure: Number; unit: events
Arm/Group | Genotype-directed, Clopidogrel | Genotype-directed, Prasugrel | Standard of Care
Number analyzed (Participants) | 5 | 0 | 4
events | 0 |  | 0

3. Secondary Outcome: Post-treatment Platelet Aggregation
Description: Platelet aggregation will be performed on a subset of subjects using VerifyNow P2Y12 which measures platelet reactivity due to the effect of a P2Y12. Values less than 180 P2Y12 Reaction Units (PRU) suggest evidence of a P2Y12 inhibitor effect. Platelet aggregation studies are optional and will not be used to modulate antiplatelet therapy.
Time Frame: 10 days
Population: Optional platelet aggregation was performed in 3 of 5 participants randomized to the Genotype-directed, clopidogrel arm and 0 of 4 participants randomized to the Standard of Care arm.
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | Genotype-directed, Clopidogrel | Genotype-directed, Prasugrel | Standard of Care
Number analyzed (Participants) | 3 | 0 | 0
percentage of inhibition | 33.7 (18.5) |  |

4. Secondary Outcome: Health Care Resource Utilization and Cost-effectiveness
Time Frame: One year
Population: This outcome measure has zero total participants analyzed because health care resource utilization and cost-effectiveness data was not collected due to the early termination of the trial.
Arm/Group | Genotype-directed, Clopidogrel | Genotype-directed, Prasugrel | Standard of Care
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Occurrence of Adverse Events
Description: The number of subjects reporting any AEs will be tabulated.
Time Frame: One year
Population: Zero participants were assigned to the genotype-directed, prasugrel group
Measure: Number; unit: participants
Arm/Group | Genotype-directed, Clopidogrel | Genotype-directed, Prasugrel | Standard of Care
Number analyzed (Participants) | 5 | 0 | 4
participants | 1 |  | 3

6. Secondary Outcome: Composite of All-cause Death, Myocardial Infarction (MI), Stroke and Repeat Revascularization
Time Frame: One year
Population: Zero participants were assigned to genotype-directed, prasugrel group
Measure: Number; unit: participants
Arm/Group | Genotype-directed, Clopidogrel | Genotype-directed, Prasugrel | Standard of Care
Number analyzed (Participants) | 5 | 0 | 4
participants | 0 |  | 0

ADVERSE EVENTS:
Time Frame: One year
Description: Zero participants were assigned to genotype-directed, prasugrel group
Arm/Group | Genotype-directed, Clopidogrel | Genotype-directed, Prasugrel | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0 | 1/4
Other Adverse Events (participants affected / at risk) | 1/5 | 0/0 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype-directed, Clopidogrel (N=5) | Genotype-directed, Prasugrel (N=0) | Standard of Care (N=4)
chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype-directed, Clopidogrel (N=5) | Genotype-directed, Prasugrel (N=0) | Standard of Care (N=4)
gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
hepatitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No